CLINICAL TRIAL: NCT05731986
Title: Neuromodulation of Blood Pressure Using Transcutaneous Spinal Stimulation in Individuals With an Acute Spinal Cord Injury - A Safety, Feasibility and Efficacy Study
Brief Title: Spinal Cord Transcutaneous Stimulation Effect on Blood Pressure in Acute Spinal Cord Injury (SCI)
Acronym: SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Einat Haber, Associate Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CSCR23FEL002; CSCR23FEL002 (Other Grant/Funding Number: New Jersey Commission on Spinal Cord Research)
Record Dates: First submitted 2023-01-25; First posted 2023-02-16 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases; Trauma, Nervous System; Nervous System Diseases; Central Nervous System Diseases; Hypotension; Orthostatic Hypotension; Cardiovascular Diseases; Acute Spinal Cord Injury; Blood Pressure
Keywords: Transcutaneous Spinal Cord Stimulation; Spinal stimulation; Orthostatic Hypotension; Blood Pressure; Neuromodulation; Acute spinal cord injury; Hypotension; Acute inpatient rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases; Trauma, Nervous System; Nervous System Diseases; Central Nervous System Diseases; Hypotension; Hypotension, Orthostatic; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Twelve individuals admitted to inpatient rehabilitation after sustaining a spinal cord injury will be enrolled. They will complete baseline assessments including an orthostatic sit-up test and neurophysiological mapping. Subsequently, the intervention will consist of two days of stimulation mapping to locate the optimal spinal segment for a blood pressure response. Participants will then be randomly assigned to two groups that would determine the order of the two testing days (optimal/sham), where stimulation is applied during an orthostatic test.
Who Masked: Participant
Masking Description: During the two testing days, participants will be blinded to the order of the stimulation. One testing day will include an orthostatic sit-up test with optimal stimulation (for a blood pressure response), while the other will include a sit-up test with sham stimulation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal stimulation (for a blood pressure response) (Active Comparator): Stimulation will be applied during an orthostatic sit-up challenge, using the profile (stimulation site and parameters) that was chosen in the mapping sessions, for optimal modulation of systolic blood pressure.
  Interventions: Diagnostic Test: Orthostatic challenge; Device: Biostim-5 transcutaneous spinal stimulation - Mapping; Device: Biostim-5 transcutaneous spinal stimulation - "Optimal" testing
- Sham stimulation (Sham Comparator): Sham stimulation will be applied during an orthostatic sit-up challenge. Sham stimulation will be delivered at a predetermined spinal location. Stimulation parameters, however, will be different from those chosen for the optimal stimulation, and sensation may be different as well.
  Interventions: Diagnostic Test: Orthostatic challenge; Device: Biostim-5 transcutaneous spinal stimulation - Mapping; Device: Biostim-5 transcutaneous spinal stimulation - "Sham" testing

INTERVENTIONS:
Diagnostic Test: Orthostatic challenge — Designed to invoke an orthostatic response. It begins with the participants lying supine on a specialized bed. The bed is then converted into a chair by raising the head of the bed by 90° and dropping the base of the bed by 90° from the knee.
  This position will be maintained for 15 minutes, while hemodynamic measures are continuously recorded. Some of these sessions will be accompanied by spinal stimulation.
  Other Names: Sit-up test
Device: Biostim-5 transcutaneous spinal stimulation - Mapping — Transcutaneous stimulation of the spinal cord. Two days of mapping will be performed to determine sites for modulation of blood pressure. During each day, with the participant in a supine or seated position, electrodes will be placed on the midline of one of the following spinous processes: C3/4, C5/6, C7/T1, T7/8, T11/12, L1/2 and S1/2. Stimulation intensity will start at 5 mA and gradually increase by 5 mA increments up to 100 mA. The frequency will be two or 30 Hz.
Device: Biostim-5 transcutaneous spinal stimulation - "Optimal" testing — Based on the mapping sessions, profiles will be established to guide the selection of an optimal site location for blood pressure modulation (within the range of 110-120 mmHg).
  Arms: Optimal stimulation (for a blood pressure response)
Device: Biostim-5 transcutaneous spinal stimulation - "Sham" testing — Based on the mapping sessions, a profile that does not elicit a significant blood pressure response, will be used for the sham stimulation.
  Arms: Sham stimulation

SUMMARY:
The goal of this clinical trial is to evaluate the effect of transcutaneous spinal cord stimulation on blood pressure in individuals with an acute spinal cord injury (within 30 days of injury). Blood pressure instability, specifically orthostatic hypotension (a drop in blood pressure when moving lying flat on your back to an upright position), appears early after the injury and often significantly interferes with participation in the critical rehabilitation time period.

The main questions it aims to answer are:

1. Can optimal spinal stimulation increase blood pressure and resolve orthostatic symptoms (such as dizziness and nausea) when individuals undergo an orthostatic provocation (a sit-up test)? Optimal stimulation and sham stimulation (which is similar to a placebo treatment) will be compared.
2. What are the various spinal sites and stimulation parameters that can be used to increase and stabilize blood pressure to the normal range of 110-120 mmHg?

Participants will undergo orthostatic tests (lying on a bed that starts out flat and then moved into an upright seated position by raising the head of bed by 90° and dropping the base of the bed by 90° from the knee) with optimal and sham stimulation, and their blood pressure measurements will be evaluated and compared.

DETAILED DESCRIPTION:
Blood pressure (BP) control in persons with a spinal cord injury (SCI) is often impaired, resulting in short and long-term health complications and a decline in quality of life. Cardiovascular (CV) dysfunction develops early after SCI and often continues a lifetime. Orthostatic hypotension (OH), a 20/10 mmHg decrease in systolic/diastolic BP when moving from a supine to an upright position, is especially prevalent in the early phase, and frequently accompanied by symptoms of dizziness, weakness, fatigue, and syncope. Affecting up to 75% of therapy treatments during inpatient rehabilitation, OH significantly interferes with participation during the critical rehab time-period, especially as length of stay in rehabilitation has substantially shortened in the past decades.

The compelling rationale for early identification and treatment of OH is met by several pharmacological and non-pharmacological interventions, however, the majority have limited effect, and increase the risk of adverse drug effects due to polypharmacy. In recent years, epidural and transcutaneous spinal cord stimulation has been explored with promising results as a potential treatment to CV dysfunction in SCI. To date, only individuals with a chronic SCI (>1 year) were included in these studies.

The objective of this study is to investigate the effect of spinal cord transcutaneous stimulation (scTS) on BP in individuals with an acute/sub-acute SCI (7-30 days after injury), during their inpatient rehabilitation. Optimal stimulation sites and parameters that increase and stabilize systolic BP (SBP) within the normotensive range (110-120 mmHg) during an orthostatic challenge will be sought. In this crossover randomized controlled trial (RCT), the effect of optimal CV stimulation and sham stimulation on BP and orthostatic symptoms will be assessed and compared.

The information gleaned from this work will allow design and implementation of scTS interventions in the early phase following an SCI, allowing full participation in inpatient rehabilitation programs, which are often hindered by the patients' autonomic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 7-30 days after injury
* Injury level ≥T2 (thoracic level)
* American Spinal Injury Association Impairment Scale (AIS) A-C
* Exhibits at least one of the following hypotensive symptoms:

  1. Baseline hypotension - resting supine or seated SBP < 90mmHg;
  2. SBP drop ≥ 20 mmHg within 5 minutes of assuming seated position;
  3. Symptoms of orthostasis with a drop of SBP (<90mmHg) from supine to sitting.

Exclusion Criteria:

* Current illness (e.g., a recent diagnosis of a deep vein thrombosis (DVT) or pulmonary embolism (PE), a pressure injury that might interfere with the intervention, etc.) or infection
* Ventilator-dependent
* History of implanted brain/spine/nerve stimulators
* Cardiac pacemaker/defibrillator or intra-cardiac lines
* Significant coronary artery or cardiac conduction disease, a recent history of myocardial infarction
* Initiated on new cardiac medications within the past 5 days
* Insufficient mental capacity to understand and independently provide consent
* Pregnancy
* Cancer
* Deemed unsuitable by study physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Optimal stimulation sites | Through Mapping and testing sessions, average of 2 weeks
  Identify scTS spinal segments that restore systolic BP within the normotensive range (110-120 mmHg).
Optimal stimulation frequency | Through Mapping and testing sessions, average of 2 weeks
  Identify scTS frequency that restores systolic BP within the normotensive range (110-120 mmHg).
Systolic blood pressure measurements (mmHg) - Mean and SD of beat-to-beat BP | Throughout the experiment, average of 2 weeks
  A comparison of systolic blood pressure with no stimulation, sham or optimal stimulation during an orthostatic challenge will be performed to assess the efficacy of stimulation.
Change in Orthostatic symptoms when stimulation is applied | Will be performed every 5 minutes during the orthostatic tests, average of 2 weeks
  A questionnaire ranking the severity of orthostatic symptoms (dizziness, nausea), using a scale of 1-10 (10 being the most severe), will be conducted during an orthostatic test to assess the efficacy of stimulation and compare the effects of optimal and sham stimulation.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) for pain | Throughout the experiment, average of 2 weeks
  Adverse effects will be recorded to assess the safety of stimulation. A numerical scale of 0 to 10 (with 10 meaning the worst pain) will be used to monitor any pain symptoms associated with the stimulation
Skin integrity assessment | Throughout the experiment, average of 2 weeks
  Adverse effects will be recorded to assess the safety of stimulation. Skin integrity (skin irritation or breakdown caused by electrodes, wires or adhesive tape) will be assessed on a daily basis
Feasibility of applying scTS in inpatient settings - compliance | Throughout the experiment, average of 2 weeks
  The ratio of total number of completed sessions divided by the number of sessions initially planned.
Feasibility of applying scTS in inpatient settings - session duration | Throughout the experiment, average of 2 weeks
  The length of time of each session and total length will be recorded.
Feasibility of applying scTS in inpatient settings - effect on therapy | Throughout the experiment, average of 2 weeks
  Total therapy time during inpatient rehabilitation will be recorded to ensure there is no interruption to the normal therapy schedule.
Electromyography (EMG) of leg muscles - muscle activation (analysis of mean and peak amplitudes) | Through Mapping and testing sessions, average of 2 weeks
  Analysis of leg-muscle EMG to identify configurations that modulate BP without eliciting motor activity, ensuring that BP response was not due to lower limb muscle contraction
Additional hemodynamic measure - diastolic blood pressure | throughout the trial, average of 2 weeks
  These measures will be collected on a daily basis throughout the trial
Additional hemodynamic measure - heart rate | throughout the trial, average of 2 weeks
  These measures will be collected on a daily basis throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Gail F Forrest, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No